CLINICAL TRIAL: NCT06770244
Title: Positive Psychology-Based Intervention Program for Postpartum Depression Within Primary Healthcare System: Protocol for a Randomized Controlled Trial
Brief Title: Positive Psychology-Based Intervention Program for Postpartum Depression Within Primary Healthcare System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yanhong Gong, Associate Professor of Social Medicne and Health Management Department, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HuazhongU20241201
Record Dates: First submitted 2025-01-06; First posted 2025-01-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Depression (PPD)
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive a positive psychology-based primary care intervention package for postpartum depression.
  Interventions: Behavioral: positive psychology-based intervention package
- Control group (No Intervention): Participants in the control group will receive usual primary care support.

INTERVENTIONS:
Behavioral: positive psychology-based intervention package — The postpartum depression intervention program will be developed in accordance with the principles of positive psychology, incorporating online psychological interventions as the primary mode of delivery. Specifically, psychological courses and training based on positive psychology will be conducted in addition to the usual community-based primary health care. Interventions use formats that include online videos and supplemental materials. The aim of the intervention is to help pregnant and postpartum women understand mental health, enhance positive emotions, improve negative emotions, maintain interpersonal relationships, and explore life meaning. Additionally, one-on-one online consultations based on positive psychology will be offered to high-risk women.
  Other Names: Holistic Well-being Intervention Framework
  Arms: Intervention group

SUMMARY:
This study is a prospective, two-arm parallel cluster randomized controlled trial that will compare the intervention effects of a positive psychology-based intervention package with usual care for postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression is one of the most common conditions affecting women during the perinatal period. It has a profound negative impact on both women's physical and mental health, manifesting in symptoms such as persistent low mood, sleep disturbances, changes in appetite, and a diminished sense of self-worth. In more severe cases, it may even lead to suicidal ideation or self-harm. Furthermore, postpartum depression significantly impairs a mother's caregiving ability, weakening the emotional bond between mother and infant. This disruption in the mother-infant relationship, in turn, can negatively affect the infant's social, emotional, and cognitive development.

Positive Psychology is an emerging subfield of psychology that focuses on the study of human positive emotions, well-being, and optimal adaptation. In contrast to traditional psychology, which primarily addresses mental illness, abnormal behaviors, and negative emotions, Positive Psychology seeks to explore and enhance the ways in which individuals and groups can thrive in areas such as positive emotions, health, and happiness. By focusing on strengths, resilience, and positive interpersonal relationships, Positive Psychology aims to foster well-being rather than merely alleviating psychological distress.

The emphasis on prevention in Positive Psychology aligns closely with the core principles of community-based primary healthcare, which prioritizes early intervention, education, and the promotion of wellness within a population. By focusing on proactive strategies that enhance mental health, Positive Psychology contributes to a broader public health agenda aimed at reducing the burden of mental disorders through early prevention rather than relying solely on treatment after the onset of illness. Therefore, integrating Positive Psychology into primary healthcare settings-particularly in the prevention and management of postpartum depression in women-offers substantial potential benefits.

This study will design a community-based intervention program for postpartum depression, centered on Positive Psychology, within the framework of the primary healthcare system. The program will be developed based on the developmental characteristics and practical needs of women experiencing postpartum depression. A cluster-randomized controlled trial will be employed to evaluate the effectiveness of the intervention. The findings will provide valuable evidence and support for mental health management measures for pregnant and postpartum women in primary healthcare settings, thereby promoting the effective implementation of maternal and child health initiatives.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* women in the early stages of pregnancy;
* adequate cognitive, comprehension, and communication abilities, and voluntary participation in the study.

Exclusion Criteria:

* individuals with severe organic or somatic diseases;
* those with a history of mental illness, substance abuse, or a family history of psychiatric disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1438 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants with postpartum depression | baseline (early pregnancy, T0), during the intervention (3 months post-randomization, T1; 6 months post-randomization, T2), and after the intervention (1 month postpartum, T3; 3 months postpartum, T4).

SECONDARY OUTCOMES:
Change in postnatal depression scale score | Baseline up to 3 months postpartum
  EPDS - Edinburgh Postnatal Depression Scale is an instrument used to measure depression. The score range is 0 to 30. A higher score means more depressed.
Anxiety Symptoms Assessment | Baseline up to 3 months postpartum
  The Generalized Anxiety Disorder 7 (GAD-7) scale is a commonly used tool for screening generalized anxiety disorder, designed to assess the severity of anxiety symptoms in participants.
Stress Assessment | Baseline up to 3 months postpartum
  The Perceived Stress Scale (PSS) primarily measures individuals' subjective perception of stress over the past month in daily life.

OTHER OUTCOMES:
Demographics Information | Baseline
  Information about the demographics of the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Community Primary Health Care Institutions, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan Z, Weng M, Su J, Yu R, Wang J, Yin X, Xia W, Gong Y. Positive psychology-based intervention programme for postpartum depression among pregnant women within the primary healthcare system: protocol for a randomised controlled trial. BMJ Open. 2025 Aug 8;15(8):e101115. doi: 10.1136/bmjopen-2025-101115. PMID 40780718